CLINICAL TRIAL: NCT06541457
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Subcutaneous Injection of HRS-7249 in Healthy Subjects - a Randomized, Double-blind, Dose-increasing, Placebo-controlled Phase I Clinical Trial
Brief Title: A Study on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-7249 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7249-101
Record Dates: First submitted 2024-07-16; First posted 2024-08-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment for intravenously: dose 1 (Experimental)
  Interventions: Drug: HRS-7249 injection; Drug: Placebo
- Treatment for intravenously: dose 2 (Experimental)
  Interventions: Drug: HRS-7249 injection; Drug: Placebo
- Treatment for intravenously: dose 3 (Experimental)
  Interventions: Drug: HRS-7249 injection; Drug: Placebo
- Treatment for intravenously: dose 4 (Experimental)
  Interventions: Drug: HRS-7249 injection; Drug: Placebo
- Treatment for intravenously: dose 5 (optional) (Experimental)
  Interventions: Drug: HRS-7249 injection; Drug: Placebo
- Treatment for intravenously: dose 6 (optional) (Experimental)
  Interventions: Drug: HRS-7249 injection; Drug: Placebo

INTERVENTIONS:
Drug: HRS-7249 injection — 6 subjects for HRS-7249 injection
Drug: Placebo — 2 subjects for placebo

SUMMARY:
It is a randomized, double-blind, single-dose, placebo-controlled phase I clinical trial. The study plans to conduct four to six dose groups of dose 1, dose 2, dose 3, dose4, dose5 (optional), and dose 6(optional). Eight subjects will be enrolled for each dose group, with six administered HRS-7249 injection and two administered placebo. A total of 32 to 48 healthy subjects are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent；
2. Age ≥ 18 and ≤ 65 years old on the day of signing the informed consent ；
3. 0.9 mmol/L≤TG≤5.6 mmol/L；
4. Male or female；
5. Male subjects weigh ≥ 50 kg and < 90 kg , female subjects weigh ≥ 45kg and < 90 kg, and BMI is in the range of 19~30 kg/m2 ；(including boundary values) Normal or abnormality such as vital signs, physical examination and laboratory examination have no clinical significance；
6. Subjects must be willing to use a highly effective method of contraception as deemed appropriate by the investigator throughout the study and for at least 6 months after the last study drug administration.

Exclusion Criteria:

1. Those who suffer from any disease that affects drug absorption, distribution, metabolism, and excretion, or can reduce compliance determined by investigators;
2. Those who suffer from any clinical diseases such as as cardiovascular, liver, kidney, digestive tract, psychiatric, hematological, metabolic abnormalities;
3. A clinically significant history of drug allergies or atopic allergic diseases (asthma, urticaria, eczematous dermatitis);
4. Those with a history of malignant diseases;
5. Those with a history of involving clinical trials of any other drugs or medical devices within the previous 3 months of screening or planned to be conducted during the study period (excluding screening failures), or those who are still within 5 half-lives of the drugs before screening (whichever is longer);
6. Those who have experienced severe trauma or surgery within the previous 6 months, or plan to undergo surgery during the trial period; Serious infected individuals within the previous 3 months of screening;
7. Those who have used any drugs during the screening period or within 2 weeks before the baseline period; or those who are still in 5 half-lives of the drug at the time of screening (whichever is longer);
8. Serum LDL-C ≥ 4.1mmol/L;
9. Platelet count<100 × 109/L;
10. Creatinine≥ upper limit of normal (ULN);
11. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma glutamyltransferase (GGT) ≥2×ULN, or total bilirubin ≥1.5×ULN;
12. During the screening period, human immunodeficiency virus antibodies (HIV-Ab), syphilis serological tests, hepatitis B virus surface antigen (HBs-Ag), or hepatitis C virus antibodies (HCV Ab) is positive;
13. Creatine kinase (CK) ≥ 3 ×ULN;
14. Thyroid stimulating hormone (TSH)< limit of normal (LLN) or≥ 1.5 ×ULN;
15. Glomerular filtration rate (eGFR)<60 mL/min/1.73m2;
16. Urine drug screening positive;
17. Those with a history of blood donation within the previous three months, severe blood loss (blood loss ≥ 400 mL), or who have received a blood transfusion within four weeks;
18. Those who have received the vaccine within the previous two weeks or plan to receive it during the trial process;
19. Those who started new physical exercise or made significantly changed their previous exercise activities within the previous 4 weeks, or who were unable to maintain basic stability in exercise during the study period;
20. Those who have made significant adjustments to their previous diet within the previous 4 weeks, or those whose diet cannot maintain basic stability during the study period;
21. Those who smoke an average of 5 or more cigarettes per day within the previous 4 weeks;
22. In the four weeks before screening, women's daily alcohol intake was more than 15 g, men's more than 25 g and more than twice a week, or the screening period and baseline period alcohol breath test (alcohol blood test can be replaced) was positive;
23. Those with a history of drug use or abuse;
24. Researchers, assistant researchers, research assistants, pharmacists, research coordinators, or other directly involved protocol implementers;
25. The researchers believe that subjects with any unfavorable factors to participate in this experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of subjects with adverse events (AEs) | Baseline up to Day 169

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: AUC0-t for HRS-7249 | Baseline up to 48 hours after dosing
  AUC0-t: Area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration
Pharmacokinetics (PK) parameter: AUC0-∞ for HRS-7249 | Baseline up to 48 hours after dosing
  AUC0-∞: Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics (PK) parameter: Cmax for HRS-7249 | Baseline up to 48 hours after dosing
  Cmax: Maximum plasma concentration
Pharmacokinetics (PK) parameter: Tmax for HRS-7249 | Baseline up to 48 hours after dosing
  Tmax: Time to reach maximum plasma concentration
Pharmacokinetics (PK) parameter: t1/2 for HRS-7249 | Baseline up to 48 hours after dosing
  t1/2: Terminal half-life
Pharmacokinetics (PK) parameter: CL/F of HRS-7249 for administration subcutaneously | Baseline up to 48 hours after dosing
  CL/F: Apparent clearance
Pharmacokinetics (PK) parameter: V/F of HRS-7249 for administration subcutaneously | Baseline up to 48 hours after dosing
  V/F: Apparent volume of distribution
Pharmacodynamics (PD): TG | Baseline up to Day 169
Pharmacodynamics (PD): HDL-C | Baseline up to Day 169
Pharmacodynamics (PD): LDL-C | Baseline up to Day 169
Pharmacodynamics (PD): non-HDL-C | Baseline up to Day 169
Pharmacodynamics (PD): VLDL-C | Baseline up to Day 169
Pharmacodynamics (PD): TC | Baseline up to Day 169
Pharmacodynamics (PD): Lp(a) | Baseline up to Day 169
Pharmacodynamics (PD): ApoB | Baseline up to Day 169
Pharmacodynamics (PD): ApoA1 | Baseline up to Day 169
Immunogenicity: Proportion of anti-drug antibodies (ADA) positive subjects | Baseline up to Day 169

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided